CLINICAL TRIAL: NCT04792970
Title: Randomized Controlled Trial of Talc Instillation In Addition To Daily Drainage Through a Tunneled Pleural Catheter to Improve Rates of Outpatient Pleurodesis in Patients With Malignant Pleural Effusion - The ASAP II Trial
Brief Title: Randomized Controlled Trial of Talc Instillation In Addition To Daily Drainage Through a Tunneled Pleural Catheter to Improve Rates of Outpatient Pleurodesis in Patients With Malignant Pleural Effusion
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study enrollment not met
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107258
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Talc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Talc instilled via tunneled pleural catheter combined with standard daily drainage (Active Comparator): This arm consists of eligible participants who are randomized to the Talc arm and would receive Talc therapy instilled into the pleural catheter.
  Interventions: Drug: Talc
- Standard daily drainage (No Intervention): This arm consists of eligible participants who are randomized to control group and would not receive any intervention.

INTERVENTIONS:
Drug: Talc — All patients randomized to the Talc arm will receive Talc therapy through the pleural catheter.
  Arms: Talc instilled via tunneled pleural catheter combined with standard daily drainage

SUMMARY:
The purpose of this study is to compare the experiences of subjects who drain malignant (cancerous) pleural effusions (fluid) from around their lung(s) in a more frequent manner using a talc instilled via tunneled pleural catheter combined with daily drainage and those subjects who drain this fluid in a daily standard manner.

DETAILED DESCRIPTION:
Study Activities: Patients will be randomized to either the standard daily drainage group or the talc instilled via tunneled pleural catheter combined with standard daily drainage group. Patients will complete questionnaires regarding their health. If you are randomized to the talc group, you will receive talc infused through the tunneled pleural catheter. If you are randomized to the standard daily drainage group, you will not receive any additional therapy. Patients will complete a drainage diary for everyday they drain fluid which will provide information on drainage volume, fluid color, pain, and complications. At 30 days and 90 days post randomization, patients will return to clinic for follow-up, at which time they will have a physical exam, chest x-ray, and complete questionnaires regarding their health.

Risks/Safety Issues: Risks associated with talc include fever and pain. Less likely risks associated with talc include infection, dyspnea, hypoxemia, pneumonia, unilateral pulmonary edema, hemoptysis, pulmonary emboli, and bronchopleural fistula.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age, inclusive.
2. Subject has a symptomatic MPE requiring intervention. For an effusion to be defined as malignant, at least one of the following must be true:

   1. There is histocytological confirmation of pleural malignancy
   2. The effusion is an exudate (per Light's criteria) in the context of histocytologically proven malignancy elsewhere, with no other clear cause for fluid identified.
3. Subject has a history of at least 1 ipsilateral pleural effusion causing dyspnea that responded to thoracentesis where the lung expanded and the dyspnea was improved.
4. Subject is willing and able to provide written informed consent.
5. Subject is willing and able to meet all study requirements, including follow-up visits and receiving study-related telephone calls.
6. Subject has sufficient pleural fluid to allow safe insertion of an IPC.
7. Subject has negative pregnancy test if appropriate.
8. Subject or caregiver is able to perform home drainage of the pleural effusion (a caregiver can be a friend, family member, or paid healthcare professional).

Exclusion Criteria:

1. Subject has significant trapped lung, or a proximal bronchial obstruction which is likely to lead to trapped lung. For a subject to be eligible for this study, two separate study center clinicians must agree that there is no significant trapped lung on the same CXR using visual estimation (reference guide). The CXR used to make this decision must have been performed ≤30 days preceding the consent form being signed, and must have been performed preferably on the same day, but no more than 7 calendar days after tunneled pleural catheter insertion. Significant trapped lung is deemed present if any 1 of the following criteria is met:

   1. A CXR shows hydropneumothorax other than small (< 1 cm between chest wall and pleural line) apical pneumothoraces.
   2. A CXR shows ≥20% of the affected hemithorax to be free of the expected lung parenchymal markings and there is no suggestion of pleural fluid.
   3. A CXR shows ≥20% of the affected hemithorax to be occupied with pleural fluid AFTER a pleural aspiration which resulted in symptoms suggestive of trapped lung (e.g., chest pain or cough).
2. Subject has a Karnofsky score <50, or a World Health Organization (WHO)/ Eastern Cooperative Oncology Group (ECOG) performance status ≥3. Subjects who have a performance status of 3 may be considered for the study if the removal of their fluid would likely improve their performance score by 1 or more.
3. Subject is pregnant, planning to become pregnant, or is lactating.
4. Subject has a history of empyema.
5. Subject has a history of chylothorax.
6. Subject has an uncorrected coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shofer, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wahidi MM, Reddy C, Yarmus L, Feller-Kopman D, Musani A, Shepherd RW, Lee H, Bechara R, Lamb C, Shofer S, Mahmood K, Michaud G, Puchalski J, Rafeq S, Cattaneo SM, Mullon J, Leh S, Mayse M, Thomas SM, Peterson B, Light RW. Randomized Trial of Pleural Fluid Drainage Frequency in Patients with Malignant Pleural Effusions. The ASAP Trial. Am J Respir Crit Care Med. 2017 Apr 15;195(8):1050-1057. doi: 10.1164/rccm.201607-1404OC. PMID 27898215
- [Background] Bhatnagar R, Keenan EK, Morley AJ, Kahan BC, Stanton AE, Haris M, Harrison RN, Mustafa RA, Bishop LJ, Ahmed L, West A, Holme J, Evison M, Munavvar M, Sivasothy P, Herre J, Cooper D, Roberts M, Guhan A, Hooper C, Walters J, Saba TS, Chakrabarti B, Gunatilake S, Psallidas I, Walker SP, Bibby AC, Smith S, Stadon LJ, Zahan-Evans NJ, Lee YCG, Harvey JE, Rahman NM, Miller RF, Maskell NA. Outpatient Talc Administration by Indwelling Pleural Catheter for Malignant Effusion. N Engl J Med. 2018 Apr 5;378(14):1313-1322. doi: 10.1056/NEJMoa1716883. PMID 29617585

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Started | 2 | 2
Completed | 1 | 1
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Undergoing Accelerated Pleurodesis
Time Frame: Up to 90 Days
Population: Only participants who underwent pleurodesis while on study are included in the analysis
Measure: Number; unit: percentage of participants
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Number analyzed (Participants) | 0 | 1
percentage of participants |  | 100

2. Secondary Outcome: Dyspnea as Measured by Questionnaire
Description: Borg Dyspnea Scale was used to rate difficulty of breathing. This scale starts at number 0 where breathing is causing no difficulty at all and progresses through to number 10 where breathing difficulty is maximal. Lower scores on this scale equal a better outcome.
Time Frame: Baseline, 30 days, 90 Days
Population: Data not collected on Standard Daily Drainage participant at day 90 due to pleurodesis at the day 30 follow-up visit.
Measure: Number; unit: score on a scale
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Number analyzed (Participants) | 1 | 1
score on a scale
  Baseline | 2 | 0.5
  Day 30 | 2 | 1
  Day 90: number analyzed (Participants) | 1 | 0
  Day 90 | 0 |

3. Secondary Outcome: Qualify of Life as Measured by Short Form 36 Health Survey (SF-36) at Baseline
Description: Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) was evaluated for overall health status. The SF-36 is composed of eight multi-item scales (Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Emotional well-being, Social functioning, Pain, General health), with scores for each of these scales (or dimensions) ranging from 0 to 100. Higher scores indicate higher qualify of life.
Time Frame: Baseline
Measure: Number; unit: score on a scale
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Number analyzed (Participants) | 1 | 1
score on a scale
  Physical functioning | 30 | 25
  Role limitations due to physical health | 0 | 0
  Role limitations due to emotional problems | 33.3 | 0
  Energy/fatigue | 50 | 25
  Emotional well-being | 56 | 72
  Social functioning | 50 | 25
  Pain | 62.5 | 0
  General health | 30 | 20

4. Secondary Outcome: Qualify of Life as Measured by Short Form 36 Health Survey (SF-36) at 30 Days
Description: as for outcome 3
Time Frame: 30 days
Measure: Number; unit: score on a scale
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Number analyzed (Participants) | 1 | 1
score on a scale
  Physical functioning | 25 | 5
  Role limitations due to physical health | 25 | 0
  Role limitations due to emotional problems | 33.3 | 0
  Energy/fatigue | 45 | 40
  Emotional well-being | 60 | 60
  Social functioning | 62.5 | 25
  Pain | 90 | 32.5
  General health | 35 | 35

5. Secondary Outcome: Qualify of Life as Measured by Short Form 36 Health Survey (SF-36) at 90 Days
Description: as for outcome 3
Time Frame: 90 days
Population: Data not collected on Standard Daily Drainage participant at day 90 due to pleurodesis at the day 30 follow-up visit.
Measure: Number; unit: score on a scale
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
Number analyzed (Participants) | 1 | 0
score on a scale
  Physical functioning | 5 |
  Role limitations due to physical health | 0 |
  Role limitations due to emotional problems | 33.3 |
  Energy/fatigue | 0 |
  Emotional well-being | 84 |
  Social functioning | 50 |
  Pain | 62.5 |
  General health | 35 |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage | Standard Daily Drainage
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 0/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage (N=2) | Standard Daily Drainage (N=2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Suspected Pleural Catheter Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Talc Instilled Via Tunneled Pleural Catheter Combined With Standard Daily Drainage (N=2) | Standard Daily Drainage (N=2)
Catheter Occlusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Worsening Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT04792970/Prot_SAP_001.pdf